CLINICAL TRIAL: NCT01400945
Title: Double Blinded, Randomized, Active Drug Comparative, Therapeutic Confirmatory Clinical Study to Evaluate the Efficacy and Safety of AGSPT201 in GERD Patients
Brief Title: Efficacy Study of AGSPT201 Tablet to Treat Gastroesophageal Reflux Disease
Acronym: AGSPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGSPT P3
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; endoscopy; LA grade; heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-Pantoprazole (Experimental): Experimental drug: AGSPT201 Tab. (contain S-Patoprazole) Active comparator: Pantoloc Tab. (contain pantoprazole)
  Interventions: Drug: AGSPT201 Tab contains S-pantoprazole

INTERVENTIONS:
Drug: AGSPT201 Tab contains S-pantoprazole — comparison of Pantoloc Tab 40mg
  Other Names: AGSPT201 Tab. (Brand name Deflux tab)

SUMMARY:
The purpose of this study is to evaluate treatment in Gastroesophageal Reflux Disease (GERD) patients (aged 18~75) with endoscopically proven GERD treated with AGSPT201 Tablet.

DETAILED DESCRIPTION:
This study is 4,8 weeks, outpatient, multicenter, randomized, double-blinded, active drug comparative, therapeutic confirmatory clinical study to evaluate the efficacy and safety of AGSPT201 in erosive esophagitis patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 18~75 years
* Patients whose esophageal lesions graded over LA A grade (The severity of lesions is classified by LA classification)
* Patients whose typical reflux symptoms such as heartburn, acid regurgitation, acid reflux and esophagus irritation during the past 3 month
* Symptoms on at least 2 days of the past 7 days

Exclusion Criteria:

* PPI treatment within 4 weeks before dosing or treatment of H2 blocker, sucralfate, prokinase NSAID (except low dose aspirin) within 2 weeks before dosing.
* Patients whose history of GI tract resection or vagotomy.
* Barrett's oesophagus greater than 3cm in length and high-grade dysplasia.
* Acid irrelevant Heartburn and regurgitation.
* Zollinger Ellison syndrome
* Hypersensitive and/or allergy to Pantoprazole and/or other PPI
* Pregnancy and lactation
* peptic ulcer
* serious hepatic
* any other renal, cardiac or haematological disease.
* Patients participated any other clinical studies during the past 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with healing of erosive esophagitis(The absence of esophageal lesions) | 4 week
  Endoscopy is performed at baseline and 4 week. All patients whose esophageal lesions are graded (LA Grade A, B, C and D). The study is completed for the patients whose esophageal lesions are healed. However patients whose esophageal lesions are not healed at 4 week were treated for an additional 4 week with endoscopy repeated at 8 week. At 8 week, the study is completed regardless healing of esophageal lesions.

SECONDARY OUTCOMES:
Absence and/or improvement of typical reflux symptoms | 4 week
  Patients recorded the improvement of typical reflux symptoms such as heartburn, acid regurgitation, acid reflux and esophagus irritation on diary card. The presence of symptoms are classified to absence (Score 0), mild (Score 1), moderate (Score 2), severe (Score 3) and very severe (Score 4).

CONTACTS AND LOCATIONS:
Overall Officials: MyoungKyu Choi, M.D, Principal Investigator — The Catholic University of Korea-St. Mary's Hospital; YoungTae Park, M.D., Study Director — Korea University Medical Center-Guro; PoongRyul Lee, M.D, Study Director — Samsung Medical Center; SangKyun Kim, M.D, Study Director — Seoul National University Hospital; HoonYong Jeong, M.D, Study Director — Asan Medical Center; SangYoung Seol, M.D, Study Director — Inje University
Locations (1):
- The Catholic University of Korea St. Mary's Hospital, Seoul, Seoul, South Korea